CLINICAL TRIAL: NCT00913523
Title: Vaginal Lactobacillus and Other Key Microflora During and After Menses in Women Using Tampons Containing Glycerol Monolaurate (GML) and Women Using Tampons Without GML
Brief Title: Clinical Evaluation of Effects of an Investigational Tampon on Vaginal Microflora
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johnson & Johnson Consumer and Personal Products Worldwide (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single
Other Study IDs: 2007-101
Record Dates: First submitted 2009-06-03; First posted 2009-06-04 (Estimated); Results first posted 2011-05-06 (Estimated); Last update posted 2011-08-23 (Estimated); Status verified 2011-08

CONDITIONS: Vaginal Microflora
Keywords: tampons; Glycerol Monolaurate; vaginal microflora; microbes; Vaginal Tampon

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Tampon with GML (Experimental): Regular and Super Tampon with GML added to the cover
  Interventions: Device: Experimental - Tampon with GML
- Tampon without GML (Sham Comparator): Regular and Super Tampon without GML
  Interventions: Device: Sham Control - Tampons without GML
- Tampon Normally Used (Sham Comparator): Type and Size of Tampon Normally Used by Subjects
  Interventions: Device: Sham Control - Tampons without GML

INTERVENTIONS:
Device: Experimental - Tampon with GML — Regular and Super Tampon with Glycerol Monolaurate (GML) added to the cover
  Other Names: Not yet marketed
  Arms: Tampon with GML
Device: Sham Control - Tampons without GML — There is no intervention associated with these arms - they are sham controls.
  Other Names: Tampons with no GML
  Arms: Tampon Normally Used; Tampon without GML

SUMMARY:
Subjects will be using investigational or control tampons during their menstrual period but these tampons are not intended to prevent, treat or diagnose an infection or other disease condition. A total 450 women will participate in this study at two study sites. Subjects will be randomly assigned to one of three tampon groups. The first group will test an experimental test tampon containing glycerol monolaurate (GML) on the cover. The second group will test an identical tampon, but without GML. The third group will not be issued study tampons but will be instructed to use their normal tampon brand. This study is intended to determine whether the effects of GML observed in the laboratory can be demonstrated in healthy menstruating women.

DETAILED DESCRIPTION:
Subjects will be using investigational or control tampons during their menstrual period but these tampons are not intended to prevent, treat or diagnose an infection or other disease condition. This study will be a randomized, single-blinded, multi-center study of women using Tampons with GML, Tampons without GML or the Tampons Normally Used for one menstrual period. Subjects will undergo Baseline microflora evaluations taken from the vaginal walls 5-10 days following their menstrual period (Baseline evaluation). Subjects will be randomly assigned to use one of the three study products during their next menstrual period. Microflora will be re-evaluated in samples taken from the tampons and from the vaginal walls during use of the study tampons, and from vaginal walls soon after the end of the menstrual period. Evaluations of microflora will be done by quantitative cultures of tampons and vaginal swabs, and also by Nugent scoring of the vaginal swabs. Staphylococcal α-hemolysin and TSST-1 will be analyzed in extracts of the study tampons from subjects found to be colonized with S. aureus. Vaginal pH will be measured, using electronic meters, at each clinic visit. All samples (tampons and vaginal swabs) will be analyzed at a central microbiology laboratory. Extracts of tampons found to contain S. aureus will be forwarded to another central laboratory for the toxin assays. Personnel in the central laboratories will be blinded to the group assignment (study product) for each subject until completion of the study.

ELIGIBILITY:
Inclusion Criteria:

* normal healthy women
* 18-45 years of age
* regular 21- to 35-day menstrual cycles with at least 5 days of bleeding, or at least 3 days of bleeding if they are using hormonal contraception
* used tampons as their principal mode of menstrual sanitary protection for at least the previous 6 months
* willing to not change their feminine care or hygiene practices during their participation in the study (except as directed by the protocol and instructions for participants)

Exclusion Criteria:

* signs or symptoms of clinically significant vulvovaginal infection or vaginosis
* history of recurrent urinary tract or vulvovaginal infection
* abnormal vaginal discharge of any etiology
* use of a systemic, vaginal, or perineal antibiotic, antifungal, anti-infective, or immunosuppressant medication or any experimental drug or medical device within the 30 days preceding the Screening/Baseline Visit
* history of treatment for Toxic Shock Syndrome (TSS) or a suspicion of having had TSS
* other clinical issues or history (per protocol) that would make participation in the trial inappropriate

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 482 (Actual)
Dates: Start 2009-01; Primary Completion 2009-08 (Actual); Study Completion 2009-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David J Chase, PhD, Study Director — Johnson & Johnson Consumer and Personal Products Worldwide
Locations (2):
- United States (2):
  - Hill Top Research, Scottsdale, Arizona
  - Hill Top Research, St. Petersburg, Florida

RESULTS

PARTICIPANT FLOW:
Groups:
- Tampon Without GML: Regular and Super Tampon without GML added to the cover
Period: Overall Study
Arm/Group | Tampon With GML | Tampon Without GML | Tampon Normally Used
Started | 162 | 159 | 161
Completed | 144 | 143 | 147
Not Completed | 18 | 16 | 14
Not completed — Withdrawal by Subject | 3 | 2 | 2
Not completed — Lost to Follow-up | 1 | 1 | 1
Not completed — Adverse Event | 1 | 0 | 0
Not completed — Protocol Violation | 5 | 8 | 8
Not completed — Pregnancy | 1 | 3 | 0
Not completed — Inadequate Number of Tampons Used | 7 | 2 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Tampon With GML | Tampon Without GML | Tampon Normally Used | Total
Number analyzed (Participants) | 162 | 159 | 161 | 482
Age, Customized [Number; unit: Participants]
  <18 years | 0 | 0 | 0 | 0
  18 to 64 years, inclusive | 162 | 159 | 161 | 482
  >=65 years | 0 | 0 | 0 | 0
Sex/Gender, Customized [Number; unit: participants]
  Female | 162 | 159 | 161 | 482
Race/Ethnicity, Customized [Number; unit: Participants]
  Hispanic or Latino (H/L) | 18 | 15 | 13 | 46
  Not Hispanic or Latino | 140 | 142 | 148 | 430
  Native Hawaiian/Other Pacific Islander (NH/OPI) | 4 | 1 | 0 | 5
  H/L & NH/OPI | 0 | 1 | 0 | 1
Race/Ethnicity, Customized [Number; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 2 | 3
  Asian | 2 | 2 | 3 | 7
  Black or African American | 17 | 12 | 21 | 50
  White | 141 | 138 | 133 | 412
  Unknown or Not Reported | 1 | 7 | 2 | 10
Region of Enrollment [Number; unit: participants]
  United States | 162 | 159 | 161 | 482
Weight 39-169 kg, inclusive [Number; unit: Participants] | 162 | 159 | 161 | 482
Height 143-148 cm, inclusive [Number; unit: Participants] | 162 | 159 | 161 | 482
Body Mass Index 15-54, inclusive [Number; unit: Participants] | 162 | 159 | 161 | 482
Average Cycle 17-35 Days, inclusive [Number; unit: Participants] — Average Days per Cycle in the past 4-6 months
  Participants | 162 | 159 | 161 | 482
Average Flow 3-10 Days, inclusive [Number; unit: Participants] — Average Days of Flow in the past 4-6 months
  Participants
    Less than 3 Days | 0 | 0 | 0 | 0
    3 to 10 Days, inclusive | 162 | 159 | 161 | 482
    More than 10 Days | 0 | 0 | 0 | 0
Number of Pregnancies Less than 14 [Number; unit: Participants] | 162 | 159 | 161 | 482
Years of Tampon Use [Number; unit: Participants]
  Less than 1 Year | 0 | 0 | 1 | 1
  1 Year | 1 | 1 | 0 | 2
  2 to 34 Years, inclusive | 161 | 158 | 160 | 479

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Subjects Showing Unfavorable Changes in Primary Microflora
Description: Percentage of subjects showing unfavorable changes of at least 1-log in lactobacilli (decrease), C. albicans (increase), or G. vaginalis (increase)
Time Frame: Mid-Cycle Baseline to Mid-Menstrual Samples
Population: Microbiological analyses are for the "per protocol" population, and no data imputation was performed. Analysis was limited to those subjects whose samples were viable for culture upon receipt at the laboratory.
Measure: Number; unit: Percentage of Participants
Arm/Group | Tampon With GML | Tampon Without GML | Tampon Normally Used
Number analyzed (Participants) | 129 | 140 | 141
Percentage of Participants | 52.7 | 52.9 | 60.0

2. Secondary Outcome: Percentage of Subjects Showing Unfavorable Changes in Primary Microflora
Description: as for outcome 1
Time Frame: Mid-Cycle Baseline to Post-Menstrual Samples
Population: as for outcome 1
Measure: Number; unit: Percentage of Participants
Arm/Group | Tampon With GML | Tampon Without GML | Tampon Normally Used
Number analyzed (Participants) | 136 | 140 | 141
Percentage of Participants | 31.6 | 34.3 | 36.4

3. Secondary Outcome: Percentage of Subjects With Selected Microflora in Tampons
Description: Percentage of subjects with selected relevant microorganisms in tampons during menses
Time Frame: During Menses
Population: as for outcome 1
Measure: Number; unit: Percentage of Participants
Arm/Group | Tampon With GML | Tampon Without GML | Tampon Normally Used
Number analyzed (Participants) | 130 | 140 | 141
Percentage of Participants
  Lactobacilli | 89.2 | 85.0 | 85.1
  C. albicans | 16.2 | 12.1 | 19.1
  G. vaginalis | 27.7 | 43.6 | 46.1
  E. coli | 28.5 | 41.4 | 34.8
  Staphylococcus aureus | 12.3 | 17.9 | 13.5
  Group B Streptococcus | 26.9 | 22.1 | 25.5
  Enterococcus sp. | 46.2 | 37.9 | 40.4

4. Secondary Outcome: Abundance of Selected Microflora in Tampons
Description: Abundance of selected relevant microorganisms in tampons during menses, in log10 colony forming units (CFU) per gram of menstrual fluid add-on to the tampon, in subjects who had detectable counts of the microorganism.
Time Frame: During Menses
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: CFU/gm
Arm/Group | Tampon With GML | Tampon Without GML | Tampon Normally Used
Number analyzed (Participants) | 130 | 140 | 141
CFU/gm
  Lactobacilli | 5.5 (1.4) | 6.0 (1.2) | 6.0 (1.2)
  C. albicans | 3.3 (1.3) | 3.7 (1.9) | 3.9 (1.5)
  G. vaginalis | 6.2 (1.5) | 6.6 (1.2) | 6.3 (1.3)
  E. coli | 4.8 (1.9) | 4.7 (2.0) | 5.1 (2.2)
  Staphylococcus aureus | 5.6 (1.9) | 4.8 (1.7) | 4.7 (1.2)
  Group B Streptococcus | 6.6 (1.7) | 6.9 (1.2) | 6.7 (1.6)
  Enterococcus sp. | 5.1 (1.5) | 5.0 (1.4) | 5.3 (1.5)

5. Secondary Outcome: Changes in Nugent Score
Description: Percentage of subjects who showed a change in Nugent score from a score of </= 3 to a score of >/= 4.
Time Frame: Mid-Cycle Baseline to Mid-Menstrual Samples
Population: as for outcome 1
Measure: Number; unit: Percentage of Participants
Arm/Group | Tampon With GML | Tampon Without GML | Tampon Normally Used
Number analyzed (Participants) | 129 | 140 | 141
Percentage of Participants | 17.7 | 19.3 | 24.8

6. Secondary Outcome: Changes in Nugent Score
Description: Percentage of subjects who showed a change in Nugent score from a score of </= 3 to a score of >/= 4.
Time Frame: Mid-Cycle Baseline to Post-Menstrual Samples
Population: as for outcome 1
Measure: Number; unit: Percentage of Participants
Arm/Group | Tampon With GML | Tampon Without GML | Tampon Normally Used
Number analyzed (Participants) | 136 | 140 | 141
Percentage of Participants | 5.9 | 12.9 | 10.6

ADVERSE EVENTS:
Time Frame: Up to 35 days
Description: One Menstrual Cycle
Arm/Group | Tampon With GML | Tampon Without GML | Tampon Normally Used
Serious Adverse Events (participants affected / at risk) | 1/162 | 3/159 | 0/161
Other Adverse Events (participants affected / at risk) | 17/162 | 17/159 | 12/161
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Tampon With GML (N=162) | Tampon Without GML (N=159) | Tampon Normally Used (N=161)
Pregnancy (Reproductive system and breast disorders) | 1 | 3 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Tampon With GML (N=162) | Tampon Without GML (N=159) | Tampon Normally Used (N=161)
Reproductive System Discomfort (Reproductive system and breast disorders) | 10 | 10 | 2 — Includes vaginal itching, dryness, irritation, odor, burning, light period, short period, heavy menstrual cramps, uterine infection, perineal irritation, groin irritation, abnormal pap smear, precancerous breast tissue, continual spotting
Upper Respiratory Discomfort (Respiratory, thoracic and mediastinal disorders) | 3 | 4 | 6 — Includes common cold, bronchitis, cough, head/sinus congestion/infection, upper respiratory infection, itching of the ears, laryngitis
Nervous System Discomfort (Nervous system disorders) | 2 | 3 | 4 — Includes headache, tension headache, anxiety, emotional stress
Dental Pain or Procedure (General disorders) | 1 | 1 | 2 — Includes tooth extraction, orthodontic pain, gum pain, dental pain
Gastrointestinal Discomfort (Gastrointestinal disorders) | 1 | 1 | 0 — Includes diarrhea and bloating
Injuries (Injury, poisoning and procedural complications) | 2 | 1 | 1 — Includes injured knee, cut ankles, muscle tension, swollen legs

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
No paper that incorporates Sponsor Confidential Information will be submitted for publication without Sponsor's prior written consent. The Institution will provide Sponsor with at least sixty (60) days for review of a manuscript, and if requested in writing, the Institution and Principal Investigators will withhold such publication for up to an additional sixty (60) days to allow for filing of a patent application.